CLINICAL TRIAL: NCT01535872
Title: Dehydroepiandrosterone Treatment for Poor Responders in IVF Patients: A Prospective Randomised Controlled Trial.
Brief Title: Study of Dehydroepiandrosterone Treatment for Poor Responders in In Vitro Fertilization Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSHFCTG34/10; SHF/CTG034/2010 (Other Grant/Funding Number: SingHealth Foundation)
Record Dates: First submitted 2012-02-15; First posted 2012-02-20 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-06

CONDITIONS: Infertility; Poor Responder to IVF Treatment
MeSH Terms: conditions — Infertility | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHEA treatment (Experimental)
  Interventions: Dietary Supplement: Dehydroepiandrosterone
- No treatment (No Intervention)

INTERVENTIONS:
Dietary Supplement: Dehydroepiandrosterone — DHEA in 25mg capsule. 1 capsule taken 3 times daily for up to 5 months.
  Arms: DHEA treatment

SUMMARY:
The aim of this study is to show solid evidences of the efficacy of DHEA in improving the success rates of in-vitro fertilization (IVF) patients facing poor ovarian reserve.

DETAILED DESCRIPTION:
Poor responders to IVF treatment occurs in 5-24% of in-vitro fertilisation (IVF) cycles, resulting in the cancellation of the cycle translating in very low pregnancy rate. Current interventions based upon the use of different stimulation regimen do not address the fundamental underlying physiological basis of follicular recruitment and development.

The over-riding objective of this proposal is to devise novel therapeutic approaches to the treatment of poor responders of IVF treatment through dietary supplementation with Dehydroepiandrosterone (DHEA). The investigators hypothesise that DHEA supplementation leads to improvements in ovarian steroidogenesis in poor responders, leading to improved IVF outcome. Specifically, the investigators aim to

1. Conduct a prospective randomised controlled trial (RCT) on the effects of DHEA supplementation in women who are poor responders to IVF treatment.
2. Investigate the effects of DHEA supplementation on ovarian steroidogenesis and biochemical and ultrasonographic markers of ovarian reserves.

ELIGIBILITY:
Inclusion Criteria:

* All women who meet one of the two following Bologna criteria for poor responder: an abnormal ovarian reserve test (AMH <1.0 ng/mL or FSH >10 IU/L ), or where fewer than 4 oocytes were retrieved or fewer than 4 follicles were observed in a previous IVF stimulation cycle with either standard long or antagonist protocols
* Where informed consent can be obtained

Exclusion Criteria:

* Previous or current DHEA supplementation
* Previous and current use of corticosteroids
* Major systemic illnesses
* Allergy to DHEA

Ages: 21 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | About one month after embryo transfer

SECONDARY OUTCOMES:
The number of oocytes retrieved at oocyte pick-up (OPU) | Within 3 weeks after ovarian stimulation
Oocyte quality | Within 3 weeks after ovarian stimulation
Number of embryos | Within 3 weeks after ovarian stimulation
Quality of embryos at the end of IVF treatment | Within 3 weeks after ovarian stimulation
The markers of ovarian reserves (AMH, follicle stimulating hormone [FSH], AFC) at the end of DHEA treatment | 4 - 5 months after DHEA treatment
Ovarian follicular levels of estradiol, testosterone, DHEA and insulin-like growth factor 1 (IGF-1) at the time of OPU | 1-2 years

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Viardot-Foucault, MD, FAMS (Endocrinology), Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore